CLINICAL TRIAL: NCT00954889
Title: Clinical Effect and Safety of Tamsulosin 0.4mg in Patients With LUTS/BPH Refractory to Tamsulosin 0.2mg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-05-004
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Tamsulosin (Experimental)
  Interventions: Drug: tamsulosin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tamsulosin — Treatment: tamsulosin 0.2mg, 2T /day Posology: two 0.2 mg tablet to be taken after an evening meal tamsulosin Tablet is an orally. (smoothly ingested without water)
  Arms: Tamsulosin
Drug: placebo — (tamsulosin 0.2mg + placebo)/day Posology: two tablet to be taken after an evening meal tamsulosin Tablet is an orally. (smoothly ingested without water)
  Arms: placebo

SUMMARY:
The purpose of this study is to explore the efficacy and safety of tamsulosin 0.4mg (Harnal® D. 0.2mg, 2T) in patients with LUTS/BPH refractory to tamsulosin 0.2mg (Harnal® D 0.2mg, 1T).

DETAILED DESCRIPTION:
Alpha-adrenoreceptor antagonists have become the primary medical treatment for lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH). The next treatment method is trans-urethral resection of prostate (TURP). TURP is the most efficient BPH treatment for relieving symptoms and improving uroflow, but it is also the invasive and morbid.

Tamsulosin has higher selectivity for the pharmacological a1-adrenoceptor subtype and the cloned a1a subtype than for the a1b subtype. Tamsulosin 0.4 mg improved Qmax to a slightly greater extent than alfuzosin 10 mg.(26% and 16% versus baseline, respectively)(http://www. fda.gov/cder/approval/ index.htm;accessed October 27, 2003.) and Tamsulosin 0.4 mg o.d. has been reported to be well tolerated irrespective of age and/or cardiovascular comorbidity/co-medication (Michel et al 1998) and no interaction with several antihypertensive agents has been reported. (Lowe et al. 1997) Our study is to explore the efficacy and safety of tamsulosin 0.4mg (Harnal® D. 0.2mg, 2T) in patients with LUTS/BPH refractory to tamsulosin 0.2mg (Harnal® D 0.2mg, 1T).

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 45years
* (LUTS/BPH patients refractory to tamsulosin 0.2mg during 4 weeks)

  *All of the following:
* Moderate to severe LUTS : IPSS ≥ 13
* An enlarged prostate (≥ 20mL, or moderately enlarged)
* Decreased peak flow rate : Qmax ≥4ml/s, ≤15mL/s volume voided ≥ 125 mL)

Exclusion Criteria:

* Post voided residual urine ≥ 200mL
* Patients performing catheterization
* Urinary tract infection patients
* Patients taking 5 alpha reductase inhibitor
* Known hypersensitivity to tamsulosin
* History of postural hypotension or syncope
* Hypertension patients treated with other alpha1-blockers
* Patients newly taking anticholinergic medication within 1 month
* Hepatic insufficiency (AST/ALT ≥ 2 times of normal range)
* Renal insufficiency (s-Cr ≥ 2mg/dL)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
To explore the efficacy of tamsulosin 0.4mg (Harnal® D. 0.2mg, 2T)in reducing the score of International Prostate Symptom Score (IPSS) from baseline to 12 weeks of treatment in patients with LUTS/BPH refractory to tamsulosin 0.2mg (Harnal® 0.2mg, 1T) | 12 weeks of treatment

SECONDARY OUTCOMES:
To evaluate efficacy on maximal flow rate and post-voided residual urine To evaluate efficacy on voiding frequency , nocturia To explore the tolerability and safety | 4 weeks and 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Lee, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Urology, Samsung Medical Center, Seoul, Seoul, South Korea